CLINICAL TRIAL: NCT04204109
Title: Interprofessional Versus Monoprofessional Case-based Learning in Childhood Cancer and the Effect on Healthcare Professionals' Interprofessional Attitudes: a Randomized Trial
Brief Title: Interprofessional Versus Monoprofessional Case-based Learning in Childhood Cancer
Acronym: INCAsE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid 19 and subsequent cancellation of all meeting activity
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Child Cancer Foundation (Other)
Responsible Party: Principal Investigator, Martha Krogh Topperzer, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Mtopperzer
Record Dates: First submitted 2019-12-10; First posted 2019-12-18 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Interprofessional Education; Continuing Professional Development; Education; Case-based Learning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interprofessional case-based learning (Experimental): The experimental intervention will be the interprofessional group receiving case-based learning about gastro-intestinal toxicities and side effects of children and adolescents with cancer.
  Interventions: Other: Interprofessional case-based learning
- Monoprofessional case-based learning (Active Comparator): The control group is the monoprofessional group that will receive the same case-based learning as the intervention group.
  Interventions: Other: Interprofessional case-based learning

INTERVENTIONS:
Other: Interprofessional case-based learning — The trial is an educational intervention where groups of healthcare professionals receive the same case-based learning: one group receives case-based learning with healthcare professionals of various professional backgrounds (experimental) versus another group receiving case-based learning with healthcare professionals exclusively of the same professional background (control).
  The educational intervention consists of a case that is developed for the purpose of the intervention.
  The participants in the experimental group will be randomised into six teams who will receive interprofessional case-based learning. The experimental group will be made up of healthcare professionals from various groups. The participants in the control group will be randomised in groups of one profession

SUMMARY:
Interprofessional education in childhood cancer is a multifaceted field. It involves multiple healthcare professionals with general and specialised knowledge and skills. Complex treatment, care and rehabilitation require continuous professional development and maintenance of healthcare professionals' competencies in their own professional field. Limited knowledge exists on comparing interprofessional and monoprofessional education and only few randomised studies have evaluated the effectiveness and efficiency of interprofessional education. One clinical area among others where healthcare professionals collaborate is in gastrointestinal toxicities and side effects. These are frequent and potentially severe clinical problems in childhood cancer that involve multiple healthcare professionals.

Objectives: To study the effect of interprofessional versus monoprofessional case-based learning on healthcare professionals' attitudes on interprofessional learning and collaboration.

Trial design: single centre investigator-initiated cluster randomized trial

Methods:

Participants: Employees with patient-related work at the childhood cancer departments and affiliated with childhood cancer at Rigshospitalet are eligible for inclusion. The setting is the childhood cancer department.

Outcome: The primary outcome is to improve healthcare professionals' interprofessional attitude.

Measurements:

The primary outcome is attitudes measured by the Assessment of Interprofessional Team Collaboration Scale (AITCS). Secondary outcome is Readiness for Interprofessional Learning Scale (RIPLS) Questionnaire, and Safety Attitudes Questionnaire (SAQ). Knowledge will be measured by written test as multiple choice questionnaire (MCQ).

Timepoints: The self-reported questionnaires will be distributed to the participants approximately one month before and one month after the educational intervention. On the day of the educational intervention, participants will answer the multiple choice questionnaire.

Analysis: Linear mixed regression will be used to compare differences in mean scores postintervention, adjusted for differences between the two groups.

Results: We hypothesise that interprofessional case-based learning positively affects the healthcare professionals' interprofessional attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals at the in-patient department for children and adolescents with cancer
* Healthcare professionals at the in-patient department for transplantation of children and adolescents with cancer
* Healthcare professionals at the out-patient departments for children and adolescents with cancer department
* Healthcare professionals affiliated with Juliane Marie Centre at Rigshospitalet
* Employees in a supportive function to the department for children and adolescents with cancer, such as psychologists, priests, pedagogues, social workers, experts in pain relief in children, physiotherapists, occupational therapists and dieticians.
* Teachers employed at a local public school but have their main working hours at the department.

Exclusion Criteria:

* Staff taking part in the intervention or in the planning of the intervention
* Management with staff responsibilities
* Lack of informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Change in the participants' interprofessional collaboration | Measured 1 month before intervention and 1-3 months after intervention in both groups
  Primary outcome: change in the participants' interprofessional attitude to collaboration measured by Assessment of interprofessional Team Collaboration Scale (AITCS). The scale contains three main categories: 1)Partnership/shared decision making (19 items), 2) Collaboration (11 items), 3) Coordination (7 items) that are rated on a scale from 1-5 (1= "never"; 2= "rarely"; 3="occasionally"; 4="most of the time"; 5="Always"). The scales procedures scores from 48 to 240. Higher scores indicate a better outcome

SECONDARY OUTCOMES:
Change in the participants' interprofessional attitudes | Measured 1 month before intervention and 1-3 months after intervention in both groups
  Secondary outcome: measured by Change in Readiness for Interprofessional Learning Survey (RIPLS). 29 items on a five-point scale 4 subscales; 1)Teamwork and collaboration, 2)Negative professional identity, 3)Positive professional identity, 4)Roles and responsibility.
  The items are rated on a scale from 1-5 (1= "strongly disagree"; 2= "agree"; 3="undecided"; 4="agree"; 5="strongly agree"). Higher scores indicate a better outcome
Change in participants' knowledge of gastrointestinal toxicities and side effects | measured at the actual intervention day 30 minutes prior to the session and immediately after the education session (maximum 15 minutes after)
  measured by written test as multiple choice questionnaire (MCQ). There are three options to chose from in this multiple choice questionnaire, one correct answer and two wrong answers. This MCQ is developed and validated for the purpose of this particular education session

CONTACTS AND LOCATIONS:
Overall Officials: Jette L Sørensen, Study Chair — Juliane Marie Centre for Women, Children and Reproduction (JMC), Rigshospitalet (RH), Copenhagen University Hospital, Denmark.
Locations (1):
- Juliane Marie Centre for Women, Children and Reproduction (JMC), Rigshospitalet (RH), Copenhagen University Hospital, Denmark., Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Randomisation is performed centrally by a computer-generated allocation sequence concealed for the investigators

REFERENCES:
- [Background] Reeves S, Pelone F, Harrison R, Goldman J, Zwarenstein M. Interprofessional collaboration to improve professional practice and healthcare outcomes. Cochrane Database Syst Rev. 2017 Jun 22;6(6):CD000072. doi: 10.1002/14651858.CD000072.pub3. PMID 28639262
- [Background] Reeves S, Zwarenstein M, Goldman J, Barr H, Freeth D, Hammick M, Koppel I. Interprofessional education: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD002213. doi: 10.1002/14651858.CD002213.pub2. PMID 18254002
- [Background] Marcussen M, Norgaard B, Borgnakke K, Arnfred S. Interprofessional clinical training in mental health improves students' readiness for interprofessional collaboration: a non-randomized intervention study. BMC Med Educ. 2019 Jan 18;19(1):27. doi: 10.1186/s12909-019-1465-6. PMID 30658648
- [Background] Ruebling I, Pole D, Breitbach AP, Frager A, Kettenbach G, Westhus N, Kienstra K, Carlson J. A comparison of student attitudes and perceptions before and after an introductory interprofessional education experience. J Interprof Care. 2014 Jan;28(1):23-7. doi: 10.3109/13561820.2013.829421. Epub 2013 Sep 3. PMID 24000881
- [Background] Norgaard B, Ammentorp J, Kofoed PE, Kyvik KO. Training improves inter-collegial communication. Clin Teach. 2012 Jun;9(3):173-7. doi: 10.1111/j.1743-498X.2011.00525.x. PMID 22587317
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Campbell MJ, Donner A, Klar N. Developments in cluster randomized trials and Statistics in Medicine. Stat Med. 2007 Jan 15;26(1):2-19. doi: 10.1002/sim.2731. PMID 17136746
- [Background] Ukoumunne OC, Gulliford MC, Chinn S, Sterne JA, Burney PG. Methods for evaluating area-wide and organisation-based interventions in health and health care: a systematic review. Health Technol Assess. 1999;3(5):iii-92. No abstract available. PMID 10982317
- [Background] Allen LM, Palermo C, Armstrong E, Hay M. Categorising the broad impacts of continuing professional development: a scoping review. Med Educ. 2019 Nov;53(11):1087-1099. doi: 10.1111/medu.13922. Epub 2019 Aug 8. PMID 31396999
- [Background] Thistlethwaite J. Interprofessional education: 50 years and counting. Med Educ. 2016 Nov;50(11):1082-1086. doi: 10.1111/medu.12959. No abstract available. PMID 27762034
- [Background] Campbell NC, Murray E, Darbyshire J, Emery J, Farmer A, Griffiths F, Guthrie B, Lester H, Wilson P, Kinmonth AL. Designing and evaluating complex interventions to improve health care. BMJ. 2007 Mar 3;334(7591):455-9. doi: 10.1136/bmj.39108.379965.BE. PMID 17332585
- [Background] Topperzer MK, Larsen HB, Hoffmann M, Schmiegelow K, Lausen B, Madsen M, Roland P, Sorensen JL. Response to: Patient-centred medical education: A proposed definition. Med Teach. 2020 Mar;42(3):360-361. doi: 10.1080/0142159X.2019.1625315. Epub 2019 Jun 12. No abstract available. PMID 31185784
- [Result] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Result] Reaman GH. Pediatric cancer research from past successes through collaboration to future transdisciplinary research. J Pediatr Oncol Nurs. 2004 May-Jun;21(3):123-7. doi: 10.1177/1043454204264406. PMID 15296038
- [Result] Christiansen HL, Bingen K, Hoag JA, Karst JS, Velazquez-Martin B, Barakat LP. Providing Children and Adolescents Opportunities for Social Interaction as a Standard of Care in Pediatric Oncology. Pediatr Blood Cancer. 2015 Dec;62 Suppl 5:S724-49. doi: 10.1002/pbc.25774. PMID 26700923
- [Result] Gatta G, Botta L, Rossi S, Aareleid T, Bielska-Lasota M, Clavel J, Dimitrova N, Jakab Z, Kaatsch P, Lacour B, Mallone S, Marcos-Gragera R, Minicozzi P, Sanchez-Perez MJ, Sant M, Santaquilani M, Stiller C, Tavilla A, Trama A, Visser O, Peris-Bonet R; EUROCARE Working Group. Childhood cancer survival in Europe 1999-2007: results of EUROCARE-5--a population-based study. Lancet Oncol. 2014 Jan;15(1):35-47. doi: 10.1016/S1470-2045(13)70548-5. Epub 2013 Dec 5. PMID 24314616
- [Result] Fish JD. No childhood cancer survivor left behind. Pediatr Blood Cancer. 2017 Feb;64(2):223-224. doi: 10.1002/pbc.26260. Epub 2016 Sep 12. No abstract available. PMID 27615193
- [Result] Schmiegelow K, Attarbaschi A, Barzilai S, Escherich G, Frandsen TL, Halsey C, Hough R, Jeha S, Kato M, Liang DC, Mikkelsen TS, Moricke A, Niinimaki R, Piette C, Putti MC, Raetz E, Silverman LB, Skinner R, Tuckuviene R, van der Sluis I, Zapotocka E; Ponte di Legno toxicity working group. Consensus definitions of 14 severe acute toxic effects for childhood lymphoblastic leukaemia treatment: a Delphi consensus. Lancet Oncol. 2016 Jun;17(6):e231-e239. doi: 10.1016/S1470-2045(16)30035-3. PMID 27299279
- [Result] Anderson RA, Marshall NS. The importance of the pediatric oncologist-nurse partnership in the delivery of total care in pediatric oncology. Med Pediatr Oncol. 2000 Apr;34(4):263-4. doi: 10.1002/(sici)1096-911x(200004)34:43.0.co;2-a. No abstract available. PMID 10742064
- [Result] Topperzer MK, Hoffmann M, Roug LI, Larsen HB, Lausen B, Schmiegelow K, Sorensen JL. Unmet need for interprofessional education in paediatric cancer: a scoping review. Support Care Cancer. 2019 Oct;27(10):3627-3637. doi: 10.1007/s00520-019-04856-4. Epub 2019 May 24. PMID 31127437
- [Result] Thomas PA, Kern DE, Hughes MT, Chen BY. Curriculum Development for Medical Education : A Six-Step Approach. Baltimore, UNITED STATES: Springer Publishing Company; 2016.
- [Result] Finley GA, Forgeron P, Arnaout M. Action research: developing a pediatric cancer pain program in jordan. J Pain Symptom Manage. 2008 Apr;35(4):447-54. doi: 10.1016/j.jpainsymman.2007.05.006. Epub 2008 Feb 6. PMID 18258410
- [Result] Lindqvist S, Duncan A, Shepstone L, Watts F, Pearce S. Case-based learning in cross-professional groups - the development of a pre-registration interprofessional learning programme. J Interprof Care. 2005 Oct;19(5):509-20. doi: 10.1080/13561820500126854. PMID 16308173
- [Result] Kiessling A, Henriksson P. Efficacy of case method learning in general practice for secondary prevention in patients with coronary artery disease: randomised controlled study. BMJ. 2002 Oct 19;325(7369):877-80. doi: 10.1136/bmj.325.7369.877. PMID 12386042
- [Result] Kiessling A, Lewitt M, Henriksson P. Case-based training of evidence-based clinical practice in primary care and decreased mortality in patients with coronary heart disease. Ann Fam Med. 2011 May-Jun;9(3):211-8. doi: 10.1370/afm.1248. PMID 21555748
- [Result] Hellman T, Jensen I, Orchard C, Bergstrom G. Preliminary testing of the Swedish version of the Assessment of Interprofessional Team Collaboration Scale (AITCS-S). J Interprof Care. 2016 Jul;30(4):499-504. doi: 10.3109/13561820.2016.1159184. Epub 2016 Jun 6. PMID 27268309
- [Result] Orchard CA, King GA, Khalili H, Bezzina MB. Assessment of Interprofessional Team Collaboration Scale (AITCS): development and testing of the instrument. J Contin Educ Health Prof. 2012 Winter;32(1):58-67. doi: 10.1002/chp.21123. PMID 22447712
- [Result] McFadyen AK, Webster V, Strachan K, Figgins E, Brown H, McKechnie J. The Readiness for Interprofessional Learning Scale: a possible more stable sub-scale model for the original version of RIPLS. J Interprof Care. 2005 Dec;19(6):595-603. doi: 10.1080/13561820500430157. PMID 16373215
- [Result] Norgaard B, Draborg E, Sorensen J. Adaptation and reliability of the Readiness for Inter professional Learning Scale in a Danish student and health professional setting. BMC Med Educ. 2016 Feb 16;16:60. doi: 10.1186/s12909-016-0591-7. PMID 26879933
- [Result] Deneckere S, Euwema M, Lodewijckx C, Panella M, Mutsvari T, Sermeus W, Vanhaecht K. Better interprofessional teamwork, higher level of organized care, and lower risk of burnout in acute health care teams using care pathways: a cluster randomized controlled trial. Med Care. 2013 Jan;51(1):99-107. doi: 10.1097/MLR.0b013e3182763312. PMID 23132203
- [Derived] Topperzer MK, Hoffmann M, Larsen HB, Rosthoj S, Nersting J, Roug LI, Pontoppidan P, Andres-Jensen L, Lausen B, Schmiegelow K, Sorensen JL. Interprofessional versus monoprofessional case-based learning in childhood cancer and the effect on healthcare professionals' knowledge and attitudes: study protocol for a randomised trial. BMC Health Serv Res. 2020 Dec 4;20(1):1124. doi: 10.1186/s12913-020-05980-2. PMID 33276789